CLINICAL TRIAL: NCT02605772
Title: A Randomized, Non-inferiority, Open-label Clinical Trial to Evaluate the Safety and Efficacy of GAcarbose+Saxagliptin Compared With Metformin+Saxagliptin in Patients With Type 2 Diabetes in Chinese
Brief Title: Safety and Efficacy of Acarbose+Saxagliptin Compared With Metformin+Saxagliptin in Patients With Type 2 Diabetes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, liao sun, principal investigator, Fifth Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FifthSunYetSen
Record Dates: First submitted 2015-11-12; First posted 2015-11-16 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Acarbose; Metformin; saxagliptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- metformin+Saxagliptin (Experimental): metformin 0.5g tablet Saxagliptin 5mg tablet metformin 0.5g three times a day for three months Saxagliptin 5mg one time a day for three months
  Interventions: Drug: Metformin; Drug: Saxagliptin
- acarbose+Saxagliptin (Experimental): acarbose 50mg tablet Saxagliptin 5mg tablet Saxagliptin 5mg one time a day for three months acarbose 100mg three times a day for three months
  Interventions: Drug: Acarbose; Drug: Saxagliptin

INTERVENTIONS:
Drug: Acarbose — group1:metformin 1.5g + Saxagliptin 5mg group2:acarbose 300mg + Saxagliptin 5mg
  Other Names: Glucobay
  Arms: acarbose+Saxagliptin
Drug: Metformin — group1:metformin 1.5g + Saxagliptin 5mg group2:acarbose 300mg + Saxagliptin 5mg
  Other Names: Glucophage
  Arms: metformin+Saxagliptin
Drug: Saxagliptin — group1:metformin 1.5g + Saxagliptin 5mg group2:acarbose 300mg + Saxagliptin 5mg
  Other Names: ONGLYZA

SUMMARY:
To investigate the Safety and Efficacy of Acarbose+Saxagliptin Compared With Metformin+Saxagliptin in Patients With Type 2 Diabetes,100 patients with T2DM will be enrolled in this study.They will randomly be assigned to Acarbose+Saxagliptin or Metformin+Saxagliptin group.HbA1c，fasting and postprandial C-peptide will be observed before and after the interventions.

DETAILED DESCRIPTION:
Participants coming on study will be assigned to two groups：Acarbose+Saxagliptin and Metformin+Saxagliptin. It may take 1 weeks to be stabilize to a standardized dose, and then the investigators will follow-up the patients for 3 months.During the period,patients will be asked to come back to the investigators center to receive the related examination every month. The investigators will detect HbA1c，fasting and postprandial C-peptide before and after the interventions.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed type 2 diabetes mellitus（course of disease less than one year） who has not receive drug treatment.
* T2DM patients who has not receive drug treatment for three months at least.
* HbA1c for 7.5-10%.

Exclusion Criteria:

* New or worsening signs or symptoms of coronary heart disease
* Medical history of active liver disease and kidney disease
* Poorly controlled hypertension（systolic blood pressure>160mmHg or diastolic blood pressure>95mmHg）
* A clinically important hematological disorder
* A history of intolerance or hypersensitivity or any contraindication to study medications (including saxagliptin, metformin, acarbose)
* Is pregnant or breast feeding or is expecting to conceive or donate eggs
* A medical history of drug abuse
* Can not be followed -up on time
* Endocrinological diseases（eg： hyperthyroidism、hypothyroidisn and cushing syndrom）
* Gastrointestinal diseases
* Mental disorser
* Hypoxic disease

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-11 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
redunction of Hemoglobin A1c (HbA1c) Levels (%) in two groups respectively after three months intervention | baseline(0 week), week twelve
  HbA1c was measured by high performance liquid chromatography with an automated biochemistry analyzer (Roche, Switzerland).

SECONDARY OUTCOMES:
Proportion of patients who achieve target of HbA1c<6.5% in two groups respectively at the end of study | baseline(0 week), week twelve
Difference of Homeostasis model assessment of insulin resistance (HOMA-IR) and Homeostasis model assessment beta cell function index (HOMA-β) between two groups after three months intervention | baseline(0 week), week twelve
  HOMA-β= Fasting C-Peptide × 0.27/(Fasting Plasma Glucose-3.5 HOMA-IR = 1.5 + Fasting Plasma Glucose × Fasting CPeptide/ 2800.